CLINICAL TRIAL: NCT01980771
Title: Barbershop Talk: HIV Prevention for African American Heterosexual Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Downstate Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Tracey Wilson, Professor, State University of New York - Downstate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5P20MD006875, subproject 5174; 5P20MD006875 (NIH)
Record Dates: First submitted 2013-10-29; First posted 2013-11-11 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: HIV
Keywords: HIV; prevention; men; African American
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Mass Screening

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BTWB intervention (Experimental): Barbershops are assigned to either experimental or active control condition. Men recruited from experimental barbershops receive a single-session group intervention focused on HIV prevention.
  Interventions: Behavioral: BTWB intervention
- Cancer prevention and screening (Active Comparator): Barbershops are assigned to either experimental or control condition. Men recruited from control barbershops receive information on cancer prevention and control.
  Interventions: Behavioral: Cancer prevention and screening

INTERVENTIONS:
Behavioral: BTWB intervention — Men work in groups to complete a intervention that takes approximately two hours to complete.
  Arms: BTWB intervention
Behavioral: Cancer prevention and screening — Men are provided health education about cancer screening and prevention
  Arms: Cancer prevention and screening

SUMMARY:
This program utilizes a community-engaged research approach to implementing and evaluating a program that seeks to reduce sexual risk behavior among Black adult heterosexual men. The investigators aims are to assess the impact of this linguistically and culturally tailored HIV prevention program on the sexual risk of heterosexual, African American men aged 18 and older, to assess the intervention's impact on the more proximal social and psychosocial variables that the program is designed to change, and to identify key contextual level factors that may impact the intervention's impact across segments of this priority population.

ELIGIBILITY:
Inclusion Criteria:

* Unprotected sex in the past three months
* Identify as Black or African American

Exclusion Criteria:

* Having been in an HIV prevention research study in the last six months
* Reporting a history in the past five years of injection drug use
* Reporting a history in the past five years of having sex with other men
* Reporting an HIV-positive serostatus
* Inability to understand spoken English.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 860 (Actual)
Dates: Start 2012-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey E Wilson, PhD, Principal Investigator — State University of New York - Downstate Medical Center
Locations (2):
- United States (2):
  - Arthur Ashe Institute for Urban Health, Inc., Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York

REFERENCES:
- [Derived] Wilson TE, Gousse Y, Joseph MA, Browne RC, Camilien B, McFarlane D, Mitchell S, Brown H, Urraca N, Romeo D, Johnson S, Salifu M, Stewart M, Vavagiakis P, Fraser M. HIV Prevention for Black Heterosexual Men: The Barbershop Talk with Brothers Cluster Randomized Trial. Am J Public Health. 2019 Aug;109(8):1131-1137. doi: 10.2105/AJPH.2019.305121. Epub 2019 Jun 20. PMID 31219715

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BTWB Intervention | Cancer Prevention and Screening
Started | 436 | 424
Completed | 352 | 305
Not Completed | 84 | 119

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BTWB Intervention | Cancer Prevention and Screening | Total
Number analyzed (Participants) | 436 | 424 | 860
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (10.8) | 34.7 (11.6) | 33.0 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 436 | 424 | 860
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 436 | 424 | 860
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 436 | 424 | 860
Living with a sexual partner [Count of Participants; unit: Participants] — Population: Missing baseline data; respondent did not answer
  Participants
    number analyzed (Participants) | 433 | 422 | 855
    (all) | 80 | 85 | 165
Current health insurance [Count of Participants; unit: Participants] — Population: Missing baseline data; respondent did not answer
  Participants
    number analyzed (Participants) | 428 | 419 | 847
    (all) | 269 | 300 | 569
Currently employed [Count of Participants; unit: Participants] — Population: Missing baseline data; respondent did not answer
  Participants
    number analyzed (Participants) | 432 | 422 | 854
    (all) | 201 | 229 | 430
High school degree or equivalent [Count of Participants; unit: Participants] — Population: Missing baseline data; respondent did not answer
  Participants
    number analyzed (Participants) | 433 | 421 | 854
    (all) | 335 | 321 | 656
Born in U.S. [Count of Participants; unit: Participants] | 233 | 324 | 557
In stable housing [Count of Participants; unit: Participants] — Population: Missing baseline data; respondent did not answer
  Participants
    number analyzed (Participants) | 431 | 423 | 854
    (all) | 363 | 290 | 653
No substance use (excludes marijuana) [Count of Participants; unit: Participants] — Population: Missing baseline data; respondent did not answer
  Participants
    number analyzed (Participants) | 433 | 424 | 857
    (all) | 392 | 351 | 743
No alcohol use [Count of Participants; unit: Participants] — Population: Missing baseline data; respondent did not answer
  Participants
    number analyzed (Participants) | 436 | 422 | 858
    (all) | 112 | 95 | 207
No incarceration history [Count of Participants; unit: Participants] — Population: Missing baseline data; respondent did not answer
  Participants
    number analyzed (Participants) | 435 | 421 | 856
    (all) | 197 | 248 | 445
No condomless sex [Count of Participants; unit: Participants] — Population: Missing baseline data; respondent did not answer
  Participants
    number analyzed (Participants) | 431 | 421 | 852
    (all) | 237 | 205 | 442

OUTCOME MEASURES:

1. Primary Outcome: Sexual Behavior
Description: Self-reported sexual behavior is the number of participants that report any unprotected anal and/or vaginal sex in the past ninety days.
Time Frame: Six month follow-up
Population: 352 men completed the six month assessment in the intervention arm; of these 347 provided complete data needed to calculate the outcome measure.
  305 men completed the six month assessment in the control arm; of these 303 provided complete data needed to calculate the outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- BTWB Intervention: Men work in groups on a single session intervention.
- Cancer Prevention and Screening: Men are provided with health education about prostate cancer screening and prevention in a single-session group format.
Arm/Group | BTWB Intervention | Cancer Prevention and Screening
Number analyzed (Participants) | 347 | 303
Participants | 225 | 163
Statistical Analysis 1: Comparison: BTWB Intervention vs Cancer Prevention and Screening; Test type: Superiority; p = 0.04, Mixed Models Analysis; Odds Ratio (OR) = 1.58, 95% CI 2-sided [1.03 to 2.43]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | BTWB Intervention | Cancer Prevention and Screening
All-Cause Mortality (participants affected / at risk) | 0/436 | 0/424
Serious Adverse Events (participants affected / at risk) | 0/436 | 0/424
Other Adverse Events (participants affected / at risk) | 2/436 | 3/424
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BTWB Intervention (N=436) | Cancer Prevention and Screening (N=424)
Incarceration (Social circumstances) | 2 (2) | 3 (3) — Participants incarcerated or at an in-patient facility as reported by contacts

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT01980771/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT01980771/SAP_001.pdf